CLINICAL TRIAL: NCT07161310
Title: A Randomized Study of Urolithin A vs. Placebo in Patients With Previously Untreated Solid Tumors Receiving Immune Checkpoint Inhibitors
Brief Title: Urolithin A in Patients With Previously Untreated Solid Tumors Receiving Immune Checkpoint Inhibitors
Acronym: MitoCancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Goethe University (Other)
Collaborators: Amazentis SA (Industry); Georg-Speyer-Haus (Unknown)
Responsible Party: Principal Investigator, Fabian Acker, Coordinating investigator, Goethe University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: Mito Cancer
Record Dates: First submitted 2025-08-22; First posted 2025-09-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Solid Cancer; Non-Small Cell Lung Cancer; Melanoma
Keywords: immune checkpoint inhibitor (ICI)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Melanoma | interventions — 3,8-dihydroxy-6H-dibenzo(b,d)pyran-6-one

STUDY DESIGN:
Intervention Model Description: A double-blinded, placebo-controlled, randomized (2:1), single-center study
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Urolithin A (Active Comparator)
  Interventions: Dietary Supplement: Urolithin A; Other: Bio specimens
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo; Other: Bio specimens

INTERVENTIONS:
Dietary Supplement: Urolithin A — Patients will receive urolithin A (UA) 1,000mg QD on from day -7 until day 60 (±7) of first-line ICI-based SACT.
  Arms: Urolithin A
Dietary Supplement: Placebo — Patients will receive placebo (PBO) on from day -7 until day 60 (±7) of first-line ICI-based SACT.
  Arms: Placebo
Other: Bio specimens — Bio specimens (PBMC, plasma, stool) will be collected during screening and on days 1, 26 (±7) and 60 (±7) of ICI.

SUMMARY:
The aim of this clinical study is to learn more about the effects of urolithin A (MitoPure®) on the immune system of cancer patients receiving immune checkpoint inhibitor-based therapies. Any effects will be compared with patients who take a placebo instead of urolithin A (MitoPure®).

ELIGIBILITY:
Inclusion Criteria:

1. Newly diagnosed solid cancer without previous systemic anticancer treatment
2. Planned single agent or double agent immune checkpoint inhibitor therapy as first-line standard-of-care treatment either with or without chemotherapy. Of note, patients receiving neoadjuvant therapy are eligible
3. Age ≥ 18 years
4. Life-expectancy ≥ 3 months
5. Eastern Cooperative Oncology Group (ECOG) Performance Status 0-1
6. Patient is willing and able to comply with the protocol for the duration of the study, including hospital visits and scheduled follow-up visits and examinations
7. Female patients of childbearing potential (WOCBP) are only eligible if using highly effective contraceptive measures and must have a negative urine or serum pregnancy test within 7 days prior to start of study treatment and must not be breast-feeding prior to start of trial. Non-child-bearing potential must be evidenced by fulfilling one of the following criteria at screening:

   * Post-menopausal defined as aged more than 50 years and amenorrheic for at least 12 months following cessation of all exogenous hormonal treatments
   * Women under 50 years old would be considered postmenopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and with LH and FSH levels in the post-menopausal range for the institution.
   * Documentation of irreversible surgical sterilization by hysterectomy, bilateral oophorectomy or bilateral salpingectomy but not tubal ligation

Exclusion Criteria:

1. Patients who currently receive or have received cytostatic chemotherapy, glucocorticoids, or immune modulatory agents (including low-dose methotrexate, TNF alpha inhibitors, calcineurin inhibitors, interleukin inhibitors, etc.) during the last 3 months are not eligible. Of note, topical glucocorticoid treatments and hormone replacement therapy is acceptable
2. Patients who currently take or plan to take mitochondrial supplements like coenzyme q10, NAD+ boosters (e.g. nicotineamide riboside, nicotineamine mononucleotide), or L-carnitine
3. Patients who have received radiotherapy to the mediastinum or to other areas with anticipated strong irradiation of a large blood vessel by the judgement of the investigator are not eligible
4. Patients with known HIV infection are not eligible. Testing is not mandatory
5. Patients with a history of solid organ or hematopoietic cell transplantation6. Any medical condition that in the opinion of the investigators would compromise the study outcome or the safety of the patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2026-01-02 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Change in the composition of circulating lymphocytes | From enrollment to the end of urolithin A intake at 8-9 weeks

SECONDARY OUTCOMES:
Changes in the plasma cytokine profile | From enrollment to the end of urolithin A intake at 8-9 weeks
Transcriptional changes in immune cells | From enrollment to the end of urolithin A intake at 8-9 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Fabian Acker, MD, Study Director — Goethe Universität
Locations (1):
- Universitätsklinikum Frankfurt, Medizinische Klinik II, Hämatologie/Onkologie, Frankfurt, Germany